CLINICAL TRIAL: NCT01004354
Title: Effect of Vitamin D Supplementation on the Metabolic Abnormalities of Second Generation Antipsychotics in Children and Adolescents
Brief Title: Vitamin D Supplementation in Psychiatric Illnesses
Acronym: VDSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Benjamin U. Nwosu, Study Principal Investigator, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Docket #13212
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Results first posted 2012-02-10 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Obesity; Vitamin D Deficiency; Psychosis; Schizophrenia; Schizoaffective Disorder
Keywords: Psychiatric illnesses; Vitamin D deficiency; Obesity
MeSH Terms: conditions — Obesity; Vitamin D Deficiency; Psychotic Disorders; Schizophrenia; Mental Disorders | interventions — Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D (Experimental)
  Interventions: Drug: Ergocalciferols

INTERVENTIONS:
Drug: Ergocalciferols — 2000 international units by mouth daily for 8 weeks.
  Other Names: Drisdol

SUMMARY:
Children and adolescents with psychiatric illnesses who are treated with medications called second generation antipsychotic agents (SGA) often gain excessive weight during their treatment with these medications. This weight gain may result in the development of features of the metabolic syndrome or frank diabetes mellitus. There is no consensus on the best way to prevent these complications. The investigators' hypothesis is that daily vitamin D supplementation in these patients will result in decreased levels of the markers of metabolic syndrome with associated reduction in waist circumference.

DETAILED DESCRIPTION:
In this 8-week open label trial, we will enroll 10 subjects who fulfill the Inclusion Criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Males/females between the ages 10 through 18 years,
2. Subjects with Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM-IV)[62] Axis 1 diagnosis who are on treatment with SGA. These conditions include schizophrenia, schizo-affective disorder, and psychosis,
3. Subjects who have gained 10% of their pre-drug body weight while receiving the following SGAs: risperidone, aripiprazole, clozapine, quetiapine and olanzapine. Subjects could be taking other psychotropic agents, but only one SGA,
4. All subjects will be able to take the prescribed vitamin D by mouth,
5. All subjects will have a 25-hydroxyvitamin D level of < 32 ng/mL,
6. All subjects must reside in an in-patient psychiatric facility.

Exclusion Criteria:

1. Pregnant or lactating women,
2. Patients with mental retardation (intelligence quotient < 50),
3. Subjects with specific systemic diseases such as diabetes mellitus, liver and kidney diseases,
4. Subjects with known history of parathyroid disorder,
5. Subjects with acquired or congenital disorders of vitamin D metabolism,
6. Subjects on calcium and vitamin D replacement therapy, such as calcium carbonate, or ergocalciferol, or cholecalciferol,
7. Subjects taking any weight loss medications, such as orlistat, and sibutramine,
8. Subjects on medications that might affect glucose levels, such as insulin or metformin.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin U Nwosu, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D: This was an open label trial that consisted of one interventional arm involving the administration of 2000 international units of ergocalciferol daily for 8 weeks.
Period: Overall Study
Arm/Group | Vitamin D
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin D
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.6 (1.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Vitamin D
Number analyzed (Participants) | 12
kilograms | 0.07 (0.06)

2. Secondary Outcome: Insulin Resistance as Measured by HOMA-IR at Baseline and Post-treatment
Description: HOMA-IR:
  It is calculated multiplying fasting plasma insulin (FPI) by fasting plasma glucose (FPG), then dividing by the constant 22.5, i.e. HOMA-IR = (FPI×FPG)/22.5
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | Vitamin D
Number analyzed (Participants) | 12
HOMA-IR score
  Baseline | 3.01 (2.65)
  Final (8 weeks) | 2.48 (2.00)

3. Secondary Outcome: Changes in Serum Levels of C-reactive Protein.
Time Frame: Baseline and 8 weeks
Population: Data were not collected for this analyte.
Arm/Group | Vitamin D
Number analyzed (Participants) | 0

4. Secondary Outcome: HDL-cholesterol at Baseline and Post-treatment
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin D
Number analyzed (Participants) | 12
mg/dL
  Baseline | 43.4 (8.75)
  Final (8 weeks) | 39.8 (9.35)

5. Secondary Outcome: LDL-cholesterol at Baseline and Post-treatment
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin D
Number analyzed (Participants) | 12
mg/dL
  Baseline | 102.00 (23.17)
  Final (8 weeks) | 86.89 (29.60)

6. Secondary Outcome: Total Cholesterol at Baseline and Post-treatment
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin D
Number analyzed (Participants) | 12
mg/dL
  Baseline | 173.67 (21.22)
  Final (8 weeks) | 161.33 (20.35)

7. Secondary Outcome: Triglycerides at Baseline and Post-treatment
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin D
Number analyzed (Participants) | 12
mg/dL
  Baseline | 189.7 (176.8)
  Final (8 weeks) | 197.9 (121.31)

8. Secondary Outcome: Adiponectin at Baseline and Post-treatment
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Vitamin D
Number analyzed (Participants) | 12
mcg/mL
  Baseline | 9.1 (4.75)
  Final (8 weeks) | 8.9 (4.7)

9. Secondary Outcome: Leptin at Baseline and Post-treatment
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D
Number analyzed (Participants) | 12
ng/mL
  Baseline | 39.23 (22.54)
  Final (8 weeks) | 43.69 (24.37)

ADVERSE EVENTS:
Arm/Group | Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No